CLINICAL TRIAL: NCT05880147
Title: App-based Consent for Participation in Pediatric Clinical Research: a Feasibility Study
Brief Title: App-based Consent for Pediatric Clinical Research
Acronym: ConsentApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Matthias Görges, PhD, Associate Professor (Partner), University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H22-01928b
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Consent
Keywords: Pediatric; Clinical research; App
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Open Label Randomized Controlled Trial
Masking Description: As blinding is impossible, we will not conceal allocation from any members of the clinical or study teams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-based consent (Experimental): Prototype consent app based on REDCap eConsent module
  Interventions: Device: Consent App
- Traditional paper-based consent (Active Comparator): Traditional paper-based consent
  Interventions: Other: Traditional paper-based consent

INTERVENTIONS:
Device: Consent App — Family will receive their study information and consent form in an app on a tablet
  Arms: App-based consent
Other: Traditional paper-based consent — Patient/family will receive their study information and consent on a traditional paper form
  Arms: Traditional paper-based consent

SUMMARY:
This study aims to understand how well app-based consent performs compared to paper-based consent when recruiting families for a clinical research project. The investigators aim to demonstrate that app-based consent is as effective as traditional methods; this will be measured by questionnaires assessing the family's comprehension and preference.

DETAILED DESCRIPTION:
Purpose and justification:

Wider access to digital technologies, familiarity with apps, and the Coronavirus disease 2019 (COVID-19) pandemic increased the demand for virtual care, prompting the need for electronic documentation of consent for research as families no longer attend in-person clinics. The investigators previously developed an app to consent patients for donating research study data in addition to traditional paper-based consent. This study aims to understand how well app-based consent performs compared to paper-based consent when recruiting families for a clinical research project.

The investigators aim to demonstrate that app-based consent is as effective as traditional methods measured by questionnaires assessing the family's comprehension and preference. If successful, this study will provide evidence for using app-based consent to enable future researchers to use similar approaches or help us further improve our app. Supporting a diverse array of consenting methods that are equivalent in promoting comprehension and participant preferences can improve research recruitment rates and increase research participant satisfaction.

Hypotheses: App-augmented consent is not inferior to traditional paper-based consent in ensuring comprehension.

Research Design:

This project will be integrated into an anesthesia study (evaluating bubble blowing as a method of distraction during IV insertions in young children, known as the BubblesRCT) by adding app-based consent and its evaluation into the regular consent flow so that families experience either app-based or traditional paper-based consent. The questions used are drawn from an established consent comprehension questionnaire and were modified to suit the requirements of our anesthesia study. Participants will also be asked a series of questions to measure characteristics like participant trust and the ease of the consenting process.

This consent modality trial will have a separate allocation schedule. Any family, who may participate in BubblesRCT, and who can be approached for consent will be allocated either to this trial's intervention (Consent modality app) or control (Consent modality paper), whereby the allocation will be switched after four participants; this is for operational feasibility purposes as randomization before approaching the parent would delay recruitment. As blinding is impossible, there will be no attempt to conceal consent modality allocation from the clinical or study teams.

Data collection:

1. The research assistant (RA) will thoroughly explain the BubblesRCT study, answer any preliminary questions, and leave the family with either a detailed paper consent form to review (Consent modality control group) or an iPad containing the consent app for review (Consent modality intervention group).
2. The family will get 15 minutes to review the consent information privately.
3. After the family have read the paper or the app-based consent form, an RA will answer any questions about the study that the family might have and invite them to consent to the BubblesRCT study. The parents will provide consent to the study either on paper or within the app (using the REDCap Electronic Informed Consent [eConsent] framework).
4. All participants who have been approached, whether the family agree to participate in the Bubbles RCT or not, will be asked to complete a comprehension questionnaire with multiple-choice questions based on a modified form of the Deaconess Informed Consent Comprehension Test (DICCT) and with a selected a set of comprehension questions with known correct answer(s) that can be used to determine accuracy.

Statistical Analysis:

The block-randomized controlled trial for non-inferiority of consent modality will tabulate results and use Wilcoxon rank sum tests for the composite comprehension correctness score. Groups will also be compared element-wise for the Likert scales using Wilcoxon rank sum tests; results may also be interpreted qualitatively.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2 to 5 years who need an IV insertion in the medical imaging department.

Exclusion Criteria:

* Children who are nonverbal;
* Children with existing vascular access
* Families who choose not to have topical anesthetic placed on their child's hands
* Children receiving anxiolytic premedication
* Children planned to undergo mask induction of anesthesia before IV placement.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of app-based consent versus paper-based consent | Immediately after consent is given for the study
  To determine better or similar comprehension of study requirements, risks and benefits, as measured by a comprehension questionnaire, and better or similar family preference for this mode of consenting. Scored using a 5-item custom multiple-choice test, with higher scores being better.

SECONDARY OUTCOMES:
Trust in the research consent process when using app-based consent versus paper-based consent | Immediately after consent is given for the study
  To determine whether app-based consent increases trust in the research consent process using a single Likert scale question (range 1-5, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Görges, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- BC Children ' s Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be presented at scientific conferences and published in peer-reviewed anesthesia journals. Once data collection is complete, a de-identified version of the data may be made available to other researchers. This is stated explicitly in the consent form, and participants are notified during the consent process that their de-identified data may be released to others for research purposes.
Supporting Information: Study Protocol, ICF
Time Frame: Once data collection is complete, de-identified data will be deposited in the University of British Columbia (UBC)'s Dataverse Repository. The study teams will keep research data for five years post-publication, as outlined in the UBC study data retention guidelines, after which it will be destroyed.
Access Criteria: Details have yet to be determined.

REFERENCES:
- [Background] Lalloo C, Pham Q, Cafazzo J, Stephenson E, Stinson J. A ResearchKit app to deliver paediatric electronic consent: Protocol of an observational study in adolescents with arthritis. Contemp Clin Trials Commun. 2020 Jan 14;17:100525. doi: 10.1016/j.conctc.2020.100525. eCollection 2020 Mar. PMID 32211557
- [Background] Blake K, Holbrook JT, Antal H, Shade D, Bunnell HT, McCahan SM, Wise RA, Pennington C, Garfinkel P, Wysocki T. Use of mobile devices and the internet for multimedia informed consent delivery and data entry in a pediatric asthma trial: Study design and rationale. Contemp Clin Trials. 2015 May;42:105-18. doi: 10.1016/j.cct.2015.03.012. Epub 2015 Apr 3. PMID 25847579
- [Background] Seltzer E, Goldshear J, Guntuku SC, Grande D, Asch DA, Klinger EV, Merchant RM. Patients' willingness to share digital health and non-health data for research: a cross-sectional study. BMC Med Inform Decis Mak. 2019 Aug 8;19(1):157. doi: 10.1186/s12911-019-0886-9. PMID 31395102
- [Background] Adjekum A, Blasimme A, Vayena E. Elements of Trust in Digital Health Systems: Scoping Review. J Med Internet Res. 2018 Dec 13;20(12):e11254. doi: 10.2196/11254. PMID 30545807
- [Background] Miller CK, O'Donnell DC, Searight HR, Barbarash RA. The Deaconess Informed Consent Comprehension Test: an assessment tool for clinical research subjects. Pharmacotherapy. 1996 Sep-Oct;16(5):872-8. PMID 8888082
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent: a new measure of understanding among research subjects. J Natl Cancer Inst. 2001 Jan 17;93(2):139-47. doi: 10.1093/jnci/93.2.139. PMID 11208884
- [Background] Sugarman J, Lavori PW, Boeger M, Cain C, Edsond R, Morrison V, Yeh SS. Evaluating the quality of informed consent. Clin Trials. 2005;2(1):34-41. doi: 10.1191/1740774505cn066oa. PMID 16279577
- See also: Pediatric Anesthesia Research Team website — https://bcchr.ca/PART